CLINICAL TRIAL: NCT02252081
Title: Dysmetabolism of Chronic Kidney Disease and Vascular Health
Brief Title: Metformin in Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENDA-014-13F; 1I01CX000982-01A1 (NIH)
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Results first posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Chronic Kidney Disease; Cardiovascular Disease; Metabolic Syndrome
Keywords: metformin; cardiovascular disease; Chronic Kidney Disease; Metabolic Syndrome
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases; Metabolic Syndrome | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- metformin (Active Comparator): 500 to 1500 mg orally per day for 16 weeks if eGFR > 45 ml/min; 500 to 1000 mg orally per day for 16 weeks if eGFR =< 45 ml/min
  Interventions: Drug: metformin
- Placebo (Placebo Comparator): placebo pill(s) orally per day for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: metformin — 500 to 1500 mg orally per day for 16 weeks if eGFR > 45 ml/min; 500 to 1000 mg orally per day for 16 weeks if eGFR =< 45 ml/min
  Arms: metformin
Drug: Placebo — placebo pill(s) orally per day for 16 weeks
  Arms: Placebo

SUMMARY:
Chronic kidney disease (CKD) is a major global health problem associated with substantial costs and resource utilization. Currently, CKD affects more than 500 million people worldwide. Patients with CKD have unacceptably high mortality rates due to cardiovascular (CV) causes, which are not entirely explained by traditional CV risk factors. The mortality rates in advanced CKD are six times higher compared to the Medicare population, with CVD accounting for the overwhelming majority of deaths. Insulin resistance (IR) is common in CKD patients and may represent a central link between CKD and the increased CVD risk observed in this population. Insulin resistance may increase CV risk by impairing and worsening endothelial function, increasing reactive oxygen species, and exacerbating systemic inflammation-hence, insulin resistance is considered a "non-traditional CV risk factor" in CKD.

Obesity (defined by a body mass index [BMI] of at least 30 kg/m2) is a major public health problem-the upward trend in obesity prevalence across regions and continents is a worldwide concern. Obesity increases the risk for cardiovascular disease and death. In the general population, obesity hastens death by 9.4 years. Obesity is an independent risk factor for CKD. Besides its contribution to the development of diabetes and hypertension, increased fat mass may also have a direct impact on kidney function.

In spite of the increasing prevalence of both obesity and CKD, the impact of obesity in the CKD population is not known, especially in terms of the exaggerated metabolic disturbances associated with their coexistence. It is highly likely that these two conditions have profound interactions that exaggerate the severity of the metabolic derangements when they coexist, particularly in regards to adipokine dysregulation, the risk of "insulin resistance", and downstream effects on vascular health. The current proposal will attempt to characterize the relative and combined impact of both obesity and CKD on metabolic disturbances, which may aid in risk stratification and identifying specific targets for intervention.

The ultimate goal of this proposal is to understand the relative and combined impact of obesity and CKD on the generation and maintenance of insulin resistance and their impact on cardiovascular health.

Specific Aim 2: To study the effects of metformin, an AMPK activator, on metabolic disturbances associated with obesity and moderate CKD.

S.A.2.a: To test if metformin will improve LAR in obese patients with moderate CKD compared to placebo.

S.A.2.b: To test if metformin will improve markers of systemic inflammation, oxidative stress, endothelial dysfunction in obese patients with moderate CKD compared to placebo.

S.A.2.c: To test if metformin will improve atherosclerosis markers and reduce clinical CVD events in obese patients with moderate CKD compared to placebo.

Hypothesis: The investigators hypothesize that the administration of metformin in obese CKD patients will significantly improve the adipokine profiles-particularly through a reduction in LAR. Additionally, that it will improve systemic inflammation, oxidative stress and endothelial function, which may or may not be mediated by changes in adipokines. Finally, the investigators hypothesize that improvements in these markers of vascular health will translate into reduced arterial stiffness and less clinical CV events

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old;
* Ability to give informed consent;
* Life expectancy greater than 6 months;
* Estimated GFR 30-59 ml/min/1.73m^2;
* Overweight (BMI >=25 to < 30 kg/m^2) or obese (BMI >=30 kg/m^2); or normal (BMI >=18.5 to <25 kg/m^2) if pre-diabetic or insulin resistant.

Exclusion Criteria:

* Pregnancy or breast feeding;
* Presence or history of Diabetes Mellitus type I or II
* History of metformin use or any insulin sensitizer or any drug for the treatment of metabolic syndrome over the last one year;
* Any acute kidney injury episode in the last 4 months due to the risk of recurrent AKI;
* Proteinuria of > 5 g in 24 hours determined by a 24 hour urine collection or PCR > 4.5;
* Uncontrolled hypertension with systolic blood pressure 160 mmHg and diastolic blood pressure 100 mmHg;
* Patients with new changes to their antihypertensive regimen over the last 1 month;
* Severe, unstable, or active inflammatory disease; active infection including seropositive HIV, Hepatitis B or C; active connective tissue disorder; or moderate to severe liver disease;
* Decompensated heart failure;
* Recent hospitalization or surgical procedure within 1 month prior to the study for any cause;
* Current active malignancy or cancer history in the prior 5 years (excluding squamous cell and basal cell skin cancers);
* Known intolerance to the study drug;
* Patient receiving oral or injected steroids
* Use of any investigational product or device within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana M Hung, MD MPH, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN
Locations (1):
- Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
No we do not plan to make individual level data available.
  This is a pilot mechanistic study.

REFERENCES:
- [Derived] El-Damanawi R, Stanley IK, Staatz C, Pascoe EM, Craig JC, Johnson DW, Mallett AJ, Hawley CM, Milanzi E, Hiemstra TF, Viecelli AK. Metformin for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2024 Jun 4;6(6):CD013414. doi: 10.1002/14651858.CD013414.pub2. PMID 38837240

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 65 patients did not meet inclusion criteria (normal GFR or to low GFR, new diabetes diagnosis, uncontrolled hypertension) or decline to participate.
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 30 | 30
Completed | 24 | 26
Not Completed | 6 | 4
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 4 | 1
Not completed — non compliance & others | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69 [64 to 72] | 66 [58 to 72] | 67 [60 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 24 | 24 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 23 | 25 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change is Leptin to Adiponectin Ratio (LAR)
Description: Change in leptin to adiponectin ratio (LAR) after 4 months of metformin vs. placebo will be assessed as a biomarker of insulin resistance in CKD
Time Frame: 16 weeks after start of treatment
Population: analyzed as log transformed using ANCOVA of change, ng/µg (log transformed value)
Measure: Median (Inter-Quartile Range); unit: ng/micrograms
Groups:
- Metformin: metformin 500 to 1500 mg orally per day for 16 weeks if eGFR > 45 ml/min/1.73m^2; 500 to 1000 mg orally per day for 16 weeks if eGFR =< 45 ml/min/1.73m^2
  Placebo: placebo pill(s) orally per day for 16 weeks
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 24 | 26
ng/micrograms
  baseline | 2.2 [1.5 to 3.2] | 1.3 [0.6 to 3.6]
  Week 16 | 1.3 [1.0 to 2.6] | 1.4 [0.5 to 3.5]

2. Secondary Outcome: Change in Flow-mediated Dilation (FMD)
Description: Change in FMD after 4 months of treatment with metformin will be compared to change in the placebo group.
Time Frame: 16 weeks after the start of treatment
Measure: Median (Inter-Quartile Range); unit: change in percent
Groups:
- Metformin: 500 to 1500 mg if eGFR > 45 ml/min; 500 to 1000 mg if eGFR =< 45 ml/min
  metformin: 500 to 1500 mg if eGFR > 45 ml/min; 500 to 1000 mg if eGFR =< 45 ml/min
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 24 | 26
change in percent
  baseline | 5.1 [3.2 to 8.4] | 5.0 [3.7 to 8.7]
  week 16 | 9.5 [5.4 to 18.8] | 6.2 [4.2 to 11.0]

3. Secondary Outcome: Aortic Pulse-wave Velocity (aPWV)
Description: is a measurement of stiffening of the large elastic arteries and atherosclerosis. It is a subclinical marker of cardiovascular disease
Time Frame: 16 weeks after starting treatment
Measure: Median (Inter-Quartile Range); unit: cm/s
Groups:
- Placebo: 500 to 1500 mg orally per day for 16 weeks if eGFR > 45 ml/min; 500 to 1000 mg orally per day for 16 weeks if eGFR =< 45 ml/min
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 24 | 26
cm/s
  baseline aPWV (cm/s) | 9.6 [8.2 to 11.4] | 9.8 [8.4 to 12.2]
  Week16 aPWC (cm/s) | 9.9 [8.9 to 10.9] | 9.9 [8.6 to 11.0]

4. Other Pre Specified Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: eGFR is a measurement of kidney function, this was a descriptive measurement
Time Frame: baseline and 16 weeks after starting treatment
Population: kidney function measurement
Measure: Median (Inter-Quartile Range); unit: ml/min
Groups:
- Metformin: metformin: 500 to 1500 mg orally per day if eGFR > 45 ml/min/1.73m^2; 500 to 1000 mg orally per day if eGFR =< 45 ml/min/1.73m^2 orally per day for 16 weeks
- Placebo: matching placebo pill(s) 500 to 1500 mg orally per day if eGFR > 45 ml/min/1.73m^2; 500 to 1000 mg orally per day if eGFR =< 45 ml/min/1.73m^2 orally per day for 16 weeks
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 24 | 26
ml/min
  baseline GFR | 49.5 [46.5 to 54.2] | 48.5 [45.4 to 56.6]
  Week 16 GFR | 52 [45.25 to 54.9] | 48.7 [43.9 to 56.5]

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: clinicaltrials.gov definitions
Arm/Group | Metformin | Placebo
All-Cause Mortality (participants affected / at risk) | 18/30 | 8/30
Serious Adverse Events (participants affected / at risk) | 2/30 | 2/30
Other Adverse Events (participants affected / at risk) | 16/30 | 6/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=30) | Placebo (N=30)
acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
pneumonia & pneumonia related complications (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pericarditis & chest pain (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=30) | Placebo (N=30)
diarrhea/loose stools/flatulence (Gastrointestinal disorders) | 8 (8) | 1 (1)
Generalized fatigue (General disorders) | 1 (1) | 1 (1)
Hyperlactetemia without acidosis >3.5 mmol/L (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — safety labs at baseline, 2,4,8,12 &16 weeks
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 2 (2)
left lower quadrant pain (Gastrointestinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT02252081/Prot_SAP_000.pdf